CLINICAL TRIAL: NCT00885833
Title: Phase I/II Study of Reduced Toxicity Myeloablative Conditioning Regimen for Wiskott-Aldrich Syndrome
Brief Title: Study of Reduced Toxicity Myeloablative Conditioning Regimen for Wiskott-Aldrich Syndrome (WAS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: The Korean Society of Hematology, The Korean Society of Pediatric Hematology Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO-S0701
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: Wiskott-Aldrich syndrome; HSCT
MeSH Terms: conditions — Wiskott-Aldrich Syndrome | interventions — fludarabine; Busulfan; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine (Experimental)
  Interventions: Drug: Fludarabine, Busulfan, Thymoglobulin

INTERVENTIONS:
Drug: Fludarabine, Busulfan, Thymoglobulin — fludarabine (40 mg/m2 once daily i.v. on days -8, -7, -6, -5, -4 & -3) busulfan (0.8 mg/kg every 6 hours i.v. on days -6, -5, -4, & -3) thymoglobulin (2.5 mg/kg once daily i.v. on days -8, -7, -6 for cord blood and on days -4, -3, -2 for bone marrow or mobilized peripheral blood)

SUMMARY:
Wiskott-Aldrich syndrome (WAS) is a rare X-linked congenital immune-deficiency syndrome and hematopoietic stem cell transplantation (HSCT) has become a curative modality. But the transplant with the conventional conditioning resulted in high incidence of treatment related toxicities and non-myeloablative conditioning resulted in high incidence of engraftment failure. Recently, fludarabine based reduced toxicity myeloablative conditioning regimen was developed for adult myeloid malignancies with promising result of good engraftment and low treatment related toxicities. To increase the engraftment potential without serious complication, reduced toxicity myeloablative conditioning regimen composed of fludarabine, busulfan, and thymoglobulin is designed for Wiskott-Aldrich syndrome.

DETAILED DESCRIPTION:
Wiskott-Aldrich syndrome (WAS) is an rare X-linked congenital immune-deficiency syndrome characterized by the triad of recurrent infection, eczema and thrombocytopenia with small size of platelet (Puck JM, 2006). Clinical studies revealed high rate of autoimmune disorder and malignancy in WAS (Ochs HD, 2006). The identification of the molecular defect in 1994 (Derry JM, 1994) has broadened the clinical spectrum of the syndrome to include chronic or intermittent X-linked thrombocytopenia (XLT), a relatively mild form of WAS and X-lined neutropenia caused by an arrest of myelopoiesis (Ochs HD, 2006).

The incidence of WAS in Korea was very low and only 6 patients diagnosed between 2001 and 2005 (Kim JG, 2006).

Conventional treatments for WAS such as prophylactic antibiotics and immune globin for infection and platelet transfusion for bleeding were not so successful (Thrasher AJ, 2000). Bone marrow transplantation (BMT) from an HLA-matched related donor is an effective treatment (Filipovich AH, 2001) and patients without appropriate related donor could receive alternative stem cell source such as matched unrelated donor or cord blood. But the transplant with the alternative donor needed more intensive conditioning to overcome the hematologic and immunologic barrier with increased treatment related toxicity. Further progress depends in particular on the development of alternative preparative conditioning regimens which allow stable engraftment of donor precursor cells with minimal systemic toxic side effects (Friedrich W, 2004).

Recently, we reported successful unrelated bone marrow transplantation in a boy with WAS with reduced toxicity myeloablative conditioning regimen to increase the engraftment potential without serious complication (Kang, 2008), and extended to multicenter phase I/II pilot study with this reduced toxicity myeloablative conditioning regimen in the HSCT for WAS.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Wiskott-Aldrich syndrome with gene analysis.
2. Indicated for hematopoietic stem cell transplantation.
3. Age: no limitation.
4. Performance status: ECOG 0-2.
5. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases:

   * Heart: a shortening fraction > 30%, ejection fraction > 45%.
   * Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
   * Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
6. Patients must lack any active viral infections or active fungal infection.
7. Appropriate hematopoietic stem cell donor is available.
8. Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant (except acute myeloid leukemia) or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2007-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the engraftment potential of fludarabine, busulfan plus thymoglobulin conditioning regimen for HSCT in WAS. | Feb. 2007 to Jan. 2012
To evaluate the incidence and severity of toxicity and treatment related mortality. | Feb. 2007 to Jan. 2012

SECONDARY OUTCOMES:
To evaluate overall and event free survival rate. | Feb. 2007 to Jan. 2012
To evaluate acute and chronic graft versus host disease (GVHD). | Feb. 2007 to Jan. 2012
To evaluate immunologic recovery after HSCT. | Feb. 2007 to Jan. 2012

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Seop Ahn, Ph. D, Principal Investigator — The Korean Society of Pediatric Hematology Oncology
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea